CLINICAL TRIAL: NCT02995928
Title: Trial of Prophylactic Decompressive Craniectomy for Poor-grade Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDSJWKDC
Record Dates: First submitted 2016-11-27; First posted 2016-12-19 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Subarachnoid Hemorrhage; Decompressive Craniectomy; Cerebral Aneurysm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm | interventions — Decompressive Craniectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompressive craniectomy (Experimental): Decompressive craniectomy and best medical treatment
  Interventions: Procedure: Decompressive craniectomy; Procedure: Best medical treatment
- Control (Active Comparator): Only best medical treatment. Decompressive craniectomy is employed only if intracranial pressure >25 mm Hg for 1-12 hours to keep the patients safe.
  Interventions: Procedure: Best medical treatment

INTERVENTIONS:
Procedure: Decompressive craniectomy — Decompressive craniectomy: All patients in the treatment group will receive decompressive craniectomy of at least 12 cm according to institutional guidelines and a published surgical protocol during the clipping surgery within 48 hours form the onset.
  Arms: Decompressive craniectomy
Procedure: Best medical treatment — Best medical treatment: Best medical treatment is based on American Heart Association/American Stroke Association (AHA/ASA) and European Stroke Organisation (ESO) as published in the current protocol from 2012 and 2013 respectively.

SUMMARY:
Decompressive craniectomy has been reported for the treatment of patients with aneurysmal subarachnoid hemorrhage (aSAH). But no prospective randomised controlled trials have yet been undertaken to confirm its effect.The purpose of the study is to determine whether decompressive craniectomy combine aneurysm clipping surgery or endovascular coiling will improve clinical outcomes of poor-grade aSAH patients.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a worldwide health burden with high fatality and permanent disability rates. Decompressive craniectomy, which is beneficial in patients with malignant middle cerebral artery infarction, may indirectly relieve the mass effect, decrease perihematomal tissue pressure, improve blood flow, reduce secondary brain damage and improve outcome without further damage to the brain due to surgery. Early therapy with either surgical clipping or neuroradiologic intervention with endovascular coiling is the primary treatment for aSAH. But whether decompressive craniectomy should be employed during the clipping surgery or immediately after coil embolization still have considerable controversy. 80 patients will be recruited to the trial over 12 months. Follow-up will take 6 months with analysis and reporting taking 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age>18yrs and age<60yrs
* It shows subarachnoid hemorrhage (SAH) based on computed tomography (CT) scan on admission
* Aneurysmal subarachnoid hemorrhage confirmed by computed tomography angiography (CTA), magnetic resonance angiography (MRA) or digital subtraction angiography (DSA)
* Presentation to our institution in World Federation of Neurological Societies (WFNS) Grade III to V neurological condition with Lateral hematoma
* Duration from onset to admission is within 48 hours

Exclusion Criteria:

* Traumatic subarachnoid hemorrhage
* Patients with cerebral herniation or highly possible to occur before surgery
* Neurosurgery contraindicated
* Patients with obvious evidence of acute hydrocephalus on admission
* Intracranial aneurysm combined with cerebral arteriovenous malformation
* Patients with obvious evidence of irreparable brainstem or thalamic injury
* Duration from onset to admission is more than 48 hours
* Disturbance of communication or poor compliance to blood collection, imageological examination and follow-up

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS) | 180 days post SAH
  By phone call following-up by senior neurosurgeons

SECONDARY OUTCOMES:
Modified Rankin scale (mRS) | 30 days and 90 days post SAH
  By phone call following-up by senior neurosurgeons
Glosgow Coma Score (GCS) | 24 hours postoperation
  Assessing by senior neurosurgeons
Incidence of delayed cerebral ischemia | 30 days post SAH
  Proved by clinical and radiologic evidence
Incidence of herniation | 30 days post SAH
  Proved by clinical and radiologic evidence
Incidence of cerebral vasospasm | 30 days post SAH
  Proved by clinical and radiologic evidence
Incidence of rebleeding | 30 days post SAH
  Proved by clinical and radiologic evidence
Death | 30 days post SAH

CONTACTS AND LOCATIONS:
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otani N, Takasato Y, Masaoka H, Hayakawa T, Yoshino Y, Yatsushige H, Miyawaki H, Sumiyoshi K, Chikashi A, Takeuchi S, Suzuki G. Surgical outcome following decompressive craniectomy for poor-grade aneurysmal subarachnoid hemorrhage in patients with associated massive intracerebral or Sylvian hematomas. Cerebrovasc Dis. 2008;26(6):612-7. doi: 10.1159/000165115. Epub 2008 Oct 23. PMID 18946217
- [Background] Uozumi Y, Sakowitz O, Orakcioglu B, Santos E, Kentar M, Haux D, Unterberg A. Decompressive craniectomy in patients with aneurysmal subarachnoid hemorrhage: a single-center matched-pair analysis. Cerebrovasc Dis. 2014;37(2):109-15. doi: 10.1159/000356979. Epub 2014 Feb 7. PMID 24514267
- [Background] Lu X, Huang B, Zheng J, Tao Y, Yu W, Tang L, Zhu R, Li S, Li L. Decompressive craniectomy for the treatment of malignant infarction of the middle cerebral artery. Sci Rep. 2014 Nov 17;4:7070. doi: 10.1038/srep07070. PMID 25400113
- [Background] Dorfer C, Frick A, Knosp E, Gruber A. Decompressive hemicraniectomy after aneurysmal subarachnoid hemorrhage. World Neurosurg. 2010 Oct-Nov;74(4-5):465-71. doi: 10.1016/j.wneu.2010.08.001. Epub 2011 Jan 12. PMID 21492596
- [Background] Schirmer CM, Hoit DA, Malek AM. Decompressive hemicraniectomy for the treatment of intractable intracranial hypertension after aneurysmal subarachnoid hemorrhage. Stroke. 2007 Mar;38(3):987-92. doi: 10.1161/01.STR.0000257962.58269.e2. Epub 2007 Feb 1. PMID 17272765
- [Background] Zhao B, Zhao Y, Tan X, Cao Y, Wu J, Zhong M, Wang S. Primary decompressive craniectomy for poor-grade middle cerebral artery aneurysms with associated intracerebral hemorrhage. Clin Neurol Neurosurg. 2015 Jun;133:1-5. doi: 10.1016/j.clineuro.2015.03.009. Epub 2015 Mar 14. PMID 25817570